CLINICAL TRIAL: NCT04888663
Title: An Open-label, Multicenter Phase Ib/II Study of Ramucirumab in Combination With Trastuzumab and Weekly Paclitaxel in Patients With HER2-positive Recurrent/Metastatic Gastric Cancer
Brief Title: Study of Ramucirumab, Trastuzumab and Paclitaxel in Patients With HER2-positive Recurrent/Metastatic Gastric Cancer (HER-RAM Study)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0275
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Recurrent/Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): (Phase Ib part) Trastuzumab 4 mg/kg (loading dose) followed by 2 mg/kg IV, ramucirumab 8 mg/kg IV, and paclitaxel 80 or 70 mg/m2 IV (according to dose level) (Phase II part) Trastuzumab 4 mg/kg (loading dose) followed by 2 mg/kg IV, ramucirumab 8 mg/kg IV, and paclitaxel at RP2D (80 or 70 mg/m2 IV)
  Interventions: Drug: Trastuzumab + Ramucirumab + Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab + Ramucirumab + Paclitaxel — For both Phase Ib and II: Trastuzumab 4 mg/kg (loading dose) followed by 2 mg/kg on Days 1, 8, 15 and 22, and ramucirumab 8 mg/kg on Days 1 and 15, as well as paclitaxel will be administered intravenously in a 4-week cycle (every 28 days) For Phase Ib, Paclitaxel 80 or 70 mg/m2 (according to dose level) will be administered on Days 1, 8, 15 For Phase II, paclitaxel at RP2D (80 or 70 mg/m2) will be administered on Days 1, 8, 15 of each cycle

SUMMARY:
Human epidermal growth factor receptor 2 (HER2) is overexpressed or amplified in 10-20% of gastric or gastroesophageal junction cancer. Trastuzumab combined with fluorouracil and platinum has been established as first-line treatment for patients with HER2-positive gastric cancer. The role of trastuzumab in second-line treatment for HER2-positive gastric cancer has not yet been addressed. Here, we evaluated the safety and efficacy of adding trastuzumab to ramucirumab and paclitaxel combination as a second-line treatment in HER2-positive gastric cancer progressed after trastuzumab-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven metastatic or locally advanced HER2-positive gastric cancer
2. Documented disease progression after receiving prior line of trastuzumab-containing chemotherapy for gastric cancer
3. Able and willing to give written informed consent and has signed the informed consent form (ICF), prior to performance of any trial activities.
4. Eligible male and female subjects aged ≥19 years.
5. Has measurable disease as determined by RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Has baseline left ventricular ejection fraction (LVEF) ≥ 55%.
8. Adequate organ function as demonstrated by laboratory test results within 14 days prior to first dose of study treatment.
9. Have urinary protein that is <2 on dipstick or routine urinalysis.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to first dose of study treatment.
11. Female subjects of childbearing potential and male subjects should be willing to use methods of birth control for the course of the study and up to 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Received prior anticancer treatment with targeted agents, chemotherapy, or radiotherapy within 14 days, with monoclonal antibodies within 28 days, has previously received treatment with ramucirumab, or has participated in another clinical trial within 14 days prior to start of study treatment.
2. Has experienced any Grade 3-4 gastrointestinal bleeding within 3 months prior to treatment.
3. Has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 3 months prior to treatment.
4. Has history of severe thromboembolism, including deep vein thrombosis and pulmonary embolism within 6 months prior to treatment.
5. Has an active or ongoing infection, symptomatic congestive heart failure, uncontrolled angina pectoris, symptomatic or poorly controlled arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator.
6. Has ongoing or active psychiatric illness or social situation that would limit compliance with study requirements.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Has evidence of active, non-infectious pneumonitis.
9. Has a known history of Human Immunodeficiency Virus (HIV).
10. Has known active hepatitis B or hepatitis C.
11. Have an elective or a planned major surgery during the course of the trial or has undergone major surgery within 4 weeks prior to enrollment.
12. Has history of GI perforation and/or fistula within 6 months prior to treatment.
13. Is pregnant or breastfeeding, or possibly pregnant.
14. Has history of Child-Pugh Class B or more of liver cirrhosis or hepatic encephalopathy, or cirrhosis with clinically meaningful ascites.
15. Is undergoing long-term antiplatelet therapy within 7 days prior to treatment.
16. Has known history of hypersensitivity to one or more of the study treatments or their substances, or known severe hypersensitivity to monoclonal antibodies.
17. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-09-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Maximum tolerated dose of trastuzumab, ramucirumab, and paclitaxel combination treatment in patients with HER2-positive gastric cancer | Phase 1b: During the first 4 weeks of treatment
Phase 2: Progression-free survival in patients with HER2-positive gastric cancer receiving trastuzumab, ramucirumab, and paclitaxel combination treatment | Phase 2: At 24 weeks after start of treatment

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 years
Objective response rate according to RECIST 1.1 | through study completion, an average of 2 years
Disease control rate according to RECIST 1.1 | through study completion, an average of 2 years
Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE v4.02 | Throughout the overall study period as well as up to 3 months after the last dose study treatment for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young RHA, MD, PhD, Principal Investigator — Yonsei Cancer Center, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CG, Jung M, Kim HS, Lee CK, Jeung HC, Koo DH, Bae WK, Zang DY, Kim BJ, Kim H, Yun UJ, Che J, Park S, Kim TS, Kwon WS, Park J, Cho SW, Nam CM, Chung HC, Rha SY. Trastuzumab Combined With Ramucirumab and Paclitaxel in Patients With Previously Treated Human Epidermal Growth Factor Receptor 2-Positive Advanced Gastric or Gastroesophageal Junction Cancer. J Clin Oncol. 2023 Sep 20;41(27):4394-4405. doi: 10.1200/JCO.22.02122. Epub 2023 Jun 26. PMID 37364218